CLINICAL TRIAL: NCT01284478
Title: Phase 2 Study of Ozurdex for Combined Pseudophakic Cystoid Macula Edema and Diabetic Macula Edema After Cataract Surgery
Brief Title: Ozurdex for Combined Pseudophakic Cystoid Macular Edema and Diabetic Macular Edema After Cataract Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northern California Retina Vitreous Associates (Other)
Collaborators: Allergan (Industry)
Responsible Party: RAHUL KHURANA, M.D. / PRINCIPAL INVESTIGATOR, NORTHERN CALIFORNIA RETINA VITREOUS ASSOCIATES
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCRVA-2011-Ozurdex-16-1
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Pseudophakic Cystoid Macular Edema,; Diabetic Macular Edema
Keywords: pseudophakic cystoid macular edema, diabetic macular edema, Irvine Gass Syndrome, cataract surgery, ozurdex, dexamethasone
MeSH Terms: conditions — Macular Edema | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexamethasone Implant (Other): Patients will be treated with the Ozurdex (Dexamethasone Implant)
  Interventions: Drug: Dexamethasone Implant

INTERVENTIONS:
Drug: Dexamethasone Implant — Ozurdex (Dexamethasone Implant), 0.7 mg will injected intravitreally

SUMMARY:
The purpose of the study is to determine where a sustained steroid delivery system (Ozurdex,Allergan) is safe and effective to treat Cystoid Macular Edema in diabetic patients after Cataract Surgery

ELIGIBILITY:
Inclusion Criteria:

* DIABETIC PATIENTS WHO DEVELOP CYSTOID MACULA EDEMA AFTER CATARACT SURGERY (WITHIN 4-10 WEEKS AFTER SURGERY
* VISUAL ACUITY WORSE THAN 20/32

Exclusion Criteria:

* VISUAL ACUITY WORSE THAN 20/200
* MODERATE OR SEVERE GLAUCOMA (AS DEFINED AS USING >2 TOPICAL GLAUCOMA MEDIATIONS.
* USE OF SYSTEMIC, PERIOCULAR OR INTRAOCULAR CORTICOSTEROIDS WITHIN 30 DAYS OF ENROLLMENT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
BEST CORRECTED VISUAL ACUITY (ETDRS) | AT DAY 180

SECONDARY OUTCOMES:
RETINAL THICKNESS MEASURED BY SPECTRAL DOMAIN OPTICAL TOMOGRAPHY | 90 and 180 DAYS
  CENTRAL FOVEAL THICKNESS AND MACULAR VOULUME

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Khurana, MD, Principal Investigator — Northern California Retina Vitreous Associates
Locations (1):
- Northern California Retina Vitreous Associates, Mountain View, California, United States